CLINICAL TRIAL: NCT03348644
Title: Milk Products in the Treatment of Hypophosphatemic Rickets: A Randomised Crossover Trial
Brief Title: Milk Products in the Treatment of Hypophosphatemic Rickets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of East Anglia (Other); Kolding Sygehus (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Milk products in HPR
Record Dates: First submitted 2017-10-09; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Hypophosphatemic Rickets
MeSH Terms: conditions — Rickets, Hypophosphatemic | interventions — Phosphates

STUDY DESIGN:
Intervention Model Description: Randomized, multiple crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phosphate tablets. (Experimental): 800 mg oral phosphor supplement distributed over five times a day independently of any prior treatment dose.
  Interventions: Dietary Supplement: Phosphate tablets.
- High cheese intake. (Active Comparator): Cheese with an estimated phosphate content of 800 mg distributed over 5 meals.
  Interventions: Dietary Supplement: High cheese intake.
- High milk intake. (Active Comparator): 800 ml of milk daily corresponding to approximately 800 mg phosphor per day.
  Interventions: Dietary Supplement: High milk intake.

INTERVENTIONS:
Dietary Supplement: Phosphate tablets.
  Arms: Phosphate tablets.
Dietary Supplement: High cheese intake.
  Arms: High cheese intake.
Dietary Supplement: High milk intake.
  Arms: High milk intake.

SUMMARY:
The aim of this study was to investigate the feasibility and efficacy of a high intake of milk and/or cheese products compared to phosphate tablets in patients with hypophosphatemic rickets when evaluating the S-phosphate levels as a main effect parameter. The study was designed as a randomized, multiple crossover study.

DETAILED DESCRIPTION:
Objectives:

Standard treatment of hypophosphatemic rickets consists of oral phosphate tablets and vitamin D analogous. Due to their rapid absorption, serum-phosphate fluctuations can occur and secondary hyperparathyroidism may be a consequence. Our aim was to evaluate, if phosphate supplement administered as milk or cheese is superior or equal to phosphate tablets in patients with hypophosphatemic rickets

Study population:

Patients with genetic verified hypophosphatemic rickets were included in the period from August 2015 to June 2016. Patients were excluded from the study if they presented with tertiary hyperparathydoism, were treated with Cinacalcet or suffered from milk allergy.

Study design:

The study was designed as a randomized, multiple crossover study with three treatment periods consisting of the regular oral phosphate supplement, a high milk intake or a high cheese intake (randomization.com). Patients were instructed to discontinue their regular treatment, except for their usual doses of D vitamin analogs, three days prior to sample collection and instead engage in the study treatment. Furthermore, they should follow their normal eating habits while undergoing the study treatment, which was controlled by food and liquid registrations.

At the phosphate supplement session, the patients were treated with an 800 mg oral phosphor supplement distributed over five times a day independently of any prior treatment dose. At the cheese session, the patients were treated with an estimated phosphate content of 800 mg distributed over 5 meals. At the milk session, the patients were treated with 800 ml of milk daily corresponding to approximately 800 mg phosphor per day.

Sampling:

After three days of treatment, the patients visited our clinic for anaerobically handled blood samples, which were collected 5 times through out one day for calcium, phosphate, parathyroid hormone, fibroblast growth factor 23 and basic phosphatase. Urine samples for calcium and phosphate was collected in containers from 0800 to 1200 and from 1200 to 1600. A 24-hour urine samples was obtained from the day before the sampling from 0800 to 0800 hours the following morning.

ELIGIBILITY:
Inclusion Criteria:

* Genetic verified hypophosphatemic rickets.
* In treated with oral phosphate tablets.

Exclusion Criteria:

* Tertiary hyperparathydoism.
* In treatment with Cinacalcet.
* Suffered from milk allergy.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Serum phosphate. | Three days.
  Evaluated in blood samples. Evaluated after three days of treatment, where we collected blood 5 times through out one day.

SECONDARY OUTCOMES:
Fibroblast growth factor 23. | Three days.
  Evaluated in blood samples. Evaluated after three days of treatment, where we collected blood 5 times through out one day.
Parathyroid hormone. | Three days.
  Evaluated in blood samples. Evaluated after three days of treatment, where we collected blood 5 times through out one day.
Total calcium. | Three days.
  Evaluated in blood samples. Evaluated after three days of treatment, where we collected blood 5 times through out one day.
Basic phosphatase. | Three days.
  Evaluated in blood samples. Evaluated after three days of treatment, where we collected blood 5 times through out one day.
Urine phosphate. | One day.
  Evaluated in urine samples. Urine samples for phosphate was collected in containers from 0800 to 1200 and from 1200 to 1600. A 24-hour urine samples was obtained from the day before the sampling from 0800 to 0800 hours the following morning.
Urine calcium. | One day.
  Evaluated in urine samples. Urine samples for calcium was collected in containers from 0800 to 1200 and from 1200 to 1600. A 24-hour urine samples was obtained from the day before the sampling from 0800 to 0800 hours the following morning.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Birkebæk., MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Publication.

REFERENCES:
- [Background] Beck-Nielsen SS, Brock-Jacobsen B, Gram J, Brixen K, Jensen TK. Incidence and prevalence of nutritional and hereditary rickets in southern Denmark. Eur J Endocrinol. 2009 Mar;160(3):491-7. doi: 10.1530/EJE-08-0818. Epub 2008 Dec 18. PMID 19095780
- [Background] Beck-Nielsen SS, Brixen K, Gram J, Brusgaard K. Mutational analysis of PHEX, FGF23, DMP1, SLC34A3 and CLCN5 in patients with hypophosphatemic rickets. J Hum Genet. 2012 Jul;57(7):453-8. doi: 10.1038/jhg.2012.56. Epub 2012 Jun 14. PMID 22695891
- [Background] Minisola S, Peacock M, Fukumoto S, Cipriani C, Pepe J, Tella SH, Collins MT. Tumour-induced osteomalacia. Nat Rev Dis Primers. 2017 Jul 13;3:17044. doi: 10.1038/nrdp.2017.44. PMID 28703220
- [Background] Bastepe M, Juppner H. Inherited hypophosphatemic disorders in children and the evolving mechanisms of phosphate regulation. Rev Endocr Metab Disord. 2008 Jun;9(2):171-80. doi: 10.1007/s11154-008-9075-3. Epub 2008 Mar 26. PMID 18365315
- [Background] Carpenter TO, Imel EA, Holm IA, Jan de Beur SM, Insogna KL. A clinician's guide to X-linked hypophosphatemia. J Bone Miner Res. 2011 Jul;26(7):1381-8. doi: 10.1002/jbmr.340. Epub 2011 May 2. PMID 21538511
- [Background] Saito H, Kusano K, Kinosaki M, Ito H, Hirata M, Segawa H, Miyamoto K, Fukushima N. Human fibroblast growth factor-23 mutants suppress Na+-dependent phosphate co-transport activity and 1alpha,25-dihydroxyvitamin D3 production. J Biol Chem. 2003 Jan 24;278(4):2206-11. doi: 10.1074/jbc.M207872200. Epub 2002 Nov 4. PMID 12419819
- [Background] Bergwitz C, Roslin NM, Tieder M, Loredo-Osti JC, Bastepe M, Abu-Zahra H, Frappier D, Burkett K, Carpenter TO, Anderson D, Garabedian M, Sermet I, Fujiwara TM, Morgan K, Tenenhouse HS, Juppner H. SLC34A3 mutations in patients with hereditary hypophosphatemic rickets with hypercalciuria predict a key role for the sodium-phosphate cotransporter NaPi-IIc in maintaining phosphate homeostasis. Am J Hum Genet. 2006 Feb;78(2):179-92. doi: 10.1086/499409. Epub 2005 Dec 9. PMID 16358214
- [Background] Nielsen LH, Rahbek ET, Beck-Nielsen SS, Christesen HT. Treatment of hypophosphataemic rickets in children remains a challenge. Dan Med J. 2014 Jul;61(7):A4874. PMID 25123121
- [Background] Peacock M, Bolognese MA, Borofsky M, Scumpia S, Sterling LR, Cheng S, Shoback D. Cinacalcet treatment of primary hyperparathyroidism: biochemical and bone densitometric outcomes in a five-year study. J Clin Endocrinol Metab. 2009 Dec;94(12):4860-7. doi: 10.1210/jc.2009-1472. Epub 2009 Oct 16. PMID 19837909
- [Background] Karp HJ, Vaihia KP, Karkkainen MU, Niemisto MJ, Lamberg-Allardt CJ. Acute effects of different phosphorus sources on calcium and bone metabolism in young women: a whole-foods approach. Calcif Tissue Int. 2007 Apr;80(4):251-8. doi: 10.1007/s00223-007-9011-7. Epub 2007 Apr 1. PMID 17401693